CLINICAL TRIAL: NCT06017063
Title: Coaching for Coping in Glioblastoma Patients and Caregivers and Its Association With Compliance to TTFields
Acronym: COCOON
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 345/2023BO1
Record Dates: First submitted 2023-07-12; First posted 2023-08-30 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-07

CONDITIONS: Compliance, Patient; Glioblastoma; Astrocytoma, Grade IV
Keywords: psychosocial support
MeSH Terms: conditions — Patient Compliance; Glioblastoma | interventions — Psychosocial Intervention

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): Patients and caregivers will participate in support program encompassing six video interventions with the BPI. Both participate in the intervention at the same time and together. The intervention starts within two weeks after start of the radiochemotherapy phase, see also figure 2. Patients and caregivers will receive an invitation link to the Vidyo sessions and can log in together to participate in the sessions.
  Interventions: Other: Psychological intervention
- Control arm (No Intervention): Patients and caregivers randomized to the control group, they will not receive the 6-week intervention by the psycho-oncologist. However, they are still entitled to guideline-based psycho-oncology counseling according to the guideline and local standard if they wish. Subsequently, they will be supported regarding coping with the disease, how to improve their mood, or which strategies are available in dealing with the disease. This conversation will last 30-60 minutes.

INTERVENTIONS:
Other: Psychological intervention — The intervention will include a psychological intervention with counseling sessions (online/video intervention) and telephone follow-up additionally to the care as usual.
  Arms: Intervention arm

SUMMARY:
The aim is to improve patients' compliance to TTFields therapy by a psychological video intervention in a multi-center, randomized controlled trial.

DETAILED DESCRIPTION:
Patients diagnosed with a glioblastoma and their family caregivers are mainly impaired by the poor prognosis and the high symptom burden. Caregivers report impaired health-related quality of life (HRQOL) and high distress. They even may experience significantly higher levels of anxiety and depression than patients themselves . Furthermore, Boele et al. showed that the overall survival in glioblastoma patients is associated with family caregivers' mastery.

In newly diagnosed glioblastoma, the EF-14 RCT demonstrated significantly prolonged survival in patients treated with TTFields compared to controls, with a median overall survival (OS) of 20.9 vs 16.0 months.

Several studies showed an important association of the daily compliance rate with OS and progression-free survival (PFS). Family caregivers' support might be associated to the patients' compliance and adequate support is required. However, so far rare supportive programs for patients and their caregivers have been established. It has been shown that delivery of supportive care via telehealth is feasible, however studies examining the effectiveness, adoption and maintenance of telehealth interventions in glioblastoma patients and family caregivers are still lacking. The aim is to improve patients' compliance to TTFields therapy by a psychological video intervention.

It is a multi-center, randomized controlled trial.

Main inclusion criteria are:

* Diagnosis of a GBM/being a GBM patient's caregiver
* Patients eligible for radiochemotherapy with TMZ and 60Gy
* Tumorboard recommendation for TTFields therapy
* Access to a computer and internet
* Absence of medical reasons precluding participation in a supportive intervention

The experimental intervention is:

Delivery of supportive care via telehealth intervention (including a brief psychological intervention and information/educational support regarding the disease, therapy and self-help options) in family caregivers and patients

The intervention encompasses six interventions (video call) for patients and caregivers.

The six sessions will be conducted by the psychologists of the coordinating center to allow homogeneous and sound implementation of the BPI. All psychologists are certified psychooncologists.

The first part of the sessions is scheduled immediately after start of radiochemotherapy (+ 2 weeks) in order to guide patients and caregivers in this important phase after first diagnose.

* First session/week 1 (+ 2 weeks) after start of radiochemotherapy: Engage and motivate patients and caregivers to participate and to develop open communication (60-90min), followed by a follow up phone call a few days later.
* Second session/week 2 (+ 2 weeks) after start of radiochemotherapy: Review of the last session and follow-up phone. Education on the techniques for optimistic attitude (including positive self-talk, positive thinking, and speaking positive). Discussion about necessity of setting achievable short-term goals in treatment process. Homework: "Write at least 3 achievable short-term goals" (45 min), followed by a follow up phone call a few days later.

The second part of the sessions is scheduled after completion of radiochemotherapy phase (+ 2 weeks) with focus in the adjuvant temozolomide therapy and TTFields therapy.

* Third session/week 7 (+ 2 weeks) after completed radiochemotherapy: Review of the last session, discussion over the phone, and homework. Providing information or advice about treatment, the TTFields therapy and medication.

  * Responding to hopelessness (focusing on positive details of the clinical course, the progress which patients made since surgery, but also sharing fears, and negative thoughts). Sharing community resources (websites, hospitals, and counseling centers).
  * Importance of TTFields therapy and association of daily compliance rate with prognosis, FAQ list, recommendations and practical aspects
  * Homework: "Provide a list of supportive resources in your community" "Provide a list of questions to the health care professionals" (45-60min), followed by a follow up phone call a few days later.
* Fourth session/week 8 (+ 2 weeks) after completed radiochemotherapy:

  * Education on the techniques for stress management (including physical activity, social contact/relationship, spending time in activity and nature (60-90 minutes) and healthy lifestyle behaviors.
  * Questions regarding TTFields and chemotherapy
  * Homework: "List the useful strategies to manage your stress during the treatment process of your partner", "Apply stress management techniques". (45-60min), followed by a follow up phone call a few days later.
* Fifth session/week 9 (+ 2 weeks) after completed radiochemotherapy:

  * First assessment after start of TTFields therapy, evaluation of practical questions and well-being
  * Education of self-care strategies (including eating well-balanced meals, permission to feel bad-schedule it in your day, permission to feel good, put off major life decisions (if it is possible), take breaks from periods of isolation, exercise - even a little bit, and let yourself cry (45-60 min).
* Sixth session/week 10 (+ 2 weeks) after completed radiochemotherapy: Feedback regarding the sessions before and planning of implementation of the learned strategies for the upcoming months. Homework: "List the strategies personally useful and what personally motivates you, learned in the last weeks"

The control condition is: Standard of care with standard access to psychosocial support in certified Neuro-Oncological Centers

Primary Outcome:

Compliance to TTFields compared in intervention and control group

Secondary Outcomes:

* Patients' health-related quality of Life (HRQoL), symptom burden, self-efficacy, anxiety, depression and its association to the intervention.
* Patient- and family caregiver-reported acceptance of intervention, patients´ acceptance of TTFields
* Adverse event of special interest: Skin irritation
* Patients' and family caregivers emotional and physical well-being,
* Correlation between endpoints to investigate dependencies of underlying concepts.
* Analysis of health utilization measures.

Optional Outcomes:

On a voluntary basis the following biosamples will be acquired for assessment of stress level and immunogenic response

* hair probes
* blood

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and give an informed consent, capacity to consent
* Given informed consent
* ≥ 18 years of age
* Patients with newly diagnosed glioblastoma
* Patients with IDH-mutant Astrocytoma, CNS WHO-Grade 4, newly diagnosed (by biopsy or incomplete tumor resection)
* Patients eligible for radiochemotherapy with temozolomide and 60 Gy
* Patients before radiochemotherapy phase or within the first 2 weeks
* Prescription of TTFields according clinical routine (including but not exclusive to)
* Access to a computer and internet
* Absence of medical reasons precluding participation in a supportive intervention

Exclusion Criteria:

* Ability to understand and give an informed consent, capacity to consent
* Given informed consent
* ≥ 18 years of age
* Being a family caregiver of a patient with newly diagnosed glioblastoma
* Access to a computer and internet
* Absence of medical reasons precluding participation in a supportive intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 275 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
EFFICACY of intervention | 9 months, last visit after completed 6 cycle of adjuvant Temozolomide (each cycle is 28 days)
  Compliance to TTFields compared in intervention and control group.Compliance will be measured by the duration of the TTFields application in each patient

SECONDARY OUTCOMES:
TOLERABILITY of psychooncological intervention | 9 months, last visit after completed 6 cycle of adjuvant Temozolomide (each cycle is 28 days)
  Patient- and caregiver-reported acceptance of intervention as measured by number of patient and cargiver dyads who completed the 6th session of the psychooncological intervention
Safety of TTFields | 9 months, last visit after completed 6 cycle of adjuvant Temozolomide (each cycle is 28 days)
  Adverse event of special interest: Skin irritation in patients under TTFields therapy
Incidence of burdened caregivers | 9 months, last visit after completed 6 cycle of adjuvant Temozolomide (each cycle is 28 days)
  Caregiver emotional and physical well-being, patient emotional and physical well-being

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol